CLINICAL TRIAL: NCT01351935
Title: Phase 1b, Escalating Dose Study of AVL-292, a Bruton's Tyrosine Kinase (Btk) Inhibitor, as Monotherapy in Subjects With Relapsed and/or Refractory B Cell Non-Hodgkin's Lymphoma, Chronic Lymphocytic Leukemia, and Waldenstrom's Macroglobulinemia
Brief Title: Escalating Dose Study in Subjects With Relapsed or Refractory B Cell Non-Hodgkin Lymphoma, Chronic Lymphocytic Leukemia, and Waldenstrom's Macroglobulinemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AVL-292-003
Record Dates: First submitted 2011-05-10; First posted 2011-05-11 (Estimated); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: B Cell Non-Hodgkin's Lymphoma; Chronic Lymphocytic Leukemia; Waldenstrom Macroglobulinemia
Keywords: non-hodgkin's lymphoma; lymphoma; leukemia; chronic lymphocytic leukemia; b-cell malignancies; Btk inhibitor; Phase 1b; Avila Therapeutics; Waldenstrom Macroglobulinemia
MeSH Terms: conditions — Lymphoma, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell; Waldenstrom Macroglobulinemia; Lymphoma, Non-Hodgkin; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AVL-292 (Experimental)
  Interventions: Drug: AVL-292

INTERVENTIONS:
Drug: AVL-292 — 125 mg to 625 mg orally, once a day, for 28 days (28 days equals 1 cycle). Number of cycles: until progression or unacceptable toxicity develops
  Other Names: Btk inhibitor

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of AVL-292 as monotherapy in subjects with relapsed or refractory B cell non-Hodgkin lymphoma (B-NHL), chronic lymphocytic leukemia (CLL) or Waldenstrom's macroglobulinemia (WM).

DETAILED DESCRIPTION:
Bruton's tyrosine kinase (Btk) is non-receptor tyrosine kinase with restricted cellular expression largely limited to B-lymphocytes, monocytes, and mast cells or basophils. Btk is a critical component of the B cell receptor (BCR) signaling network and is crucial for B cell development. Investigation has revealed that some B cell lymphomas and CLL depend on BCR signaling, suggesting that interruption of such signaling could be a promising therapeutic opportunity in B-NHL, CLL and WM.

ELIGIBILITY:
Inclusion Criteria:

* Women and men ≥18 years of age
* Body weight ≥50 kg.
* Confirmed diagnosis of B cellNon-Hodgkin Lymphoma(according to World Health Organization [WHO] classification)including Chronic Lymphocytic Leukemia/Small cell Lymphocytic Leukemia (International Workshop),or Waldenstrom's Macroglobulinemia(Second International Workshop)
* Have failed ≥1 previous treatment for B-NHL/CLL/WM, and have relapsed or refractory disease following last prior treatment.
* Eastern Cooperative Oncology Group performance status of ≤ 2 and a life expectancy of at least 3 months.
* Ability to swallow oral capsules without difficulty
* Has recovered from adverse toxic effects of prior therapies
* Meet the following clinical laboratory requirements:

  * Creatinine ≤ 1.5 × upper limit of normal (ULN)
  * Total bilirubin ≤ 1.5 x ULN
  * AST and ALT ≤ 3 × ULN
  * Platelet count ≥ 50,000/µL (non-hodgkin & Waldenstrom's)
  * Platelet count ≥ 30,000/µL (chronic lymphocytic leukemia)
  * Absolute Neutrophil count ≥ 1000/µL

Exclusion Criteria:

* Prior allogeneic bone marrow transplant
* Autologous stem cell transplant within 3 months of screening
* Active central nervous system involvement
* Subjects with autoimmune hemolytic anemia or immune thrombocytopenia
* Prior treatment with a Btk inhibitor
* Active uncontrolled infection
* History of malabsorption
* Uncontrolled illness, i.e cardiac, endocrine, respiratory, etc.
* History of myocardial infarction, acute coronary syndromes, coronary angioplasty and/or stenting with in the previous 6 months
* History of another currently active cancer
* History of major surgery within 4 weeks or minor surgery within 1 week
* Other medical or psychiatric illness or organ dysfunction
* HIV positive
* Positive for Hepatitis B surface antigen or Hepatitis C-virus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2011-07-18 (Actual); Primary Completion 2015-06-26 (Actual); Study Completion 2015-06-26 (Actual)

PRIMARY OUTCOMES:
Safety, tolerability,and dose limiting toxicities will be determined using AEs,PE,ophthalmologic examinations,clinical laboratory tests,vital signs, ECGs and echocardiograms/MUGA scans. | with in the first 28 days after initiation of once daily oral dosing

SECONDARY OUTCOMES:
Establish recommended Phase 2 dose, after completing dose escalation in Part 1 and evaluating accumulated safety,PK,and PD data from the dose escalation phase (Part1) | Completion of Part 1 dose escalation phase of study
  After completion of observation for dose limiting toxicities in Part 1 of the study, the accumulated safety, PK, and PD data from Part 1 will be evaluated by the investigators and Sponsor to select a preliminary RP2D for administration to additional subjects to be enrolled into 1 of 3 independent and non-randomized diagnosis-specific expansion cohorts in Part 2 of the study
Evaluate the Pharmacokinetic parameters of AVL-292 | First 28 days of dosing
  Serial blood sampling to enable PK characterization of AVL-292 will be performed for the Cycle1 Day 1 (C1D1) and Cycle 1Day 15 dose administrations. Additional samples will be obtained on C1D8 and C1D22.A non-compartmental model will be evaluated for all subjects.
Evaluate the Pharmacodynamics of AVL-292 by measurement of free Btk | First 28 days of dosing
  The PD activity of AVL-292 will be studied with a quantitative assay using a covalent probe to directly assess free Btk in PBMC lysates.
Characterize preliminary anti-tumor efficacy of AVL-292 in relapsed and/or refractory B-NHL, CLL and WM | After completion of 28 day cycle of treatment
  Efficacy response assessments will be formally assessed within 7 days preceding C2D1, C3D1, C5D1, C7D1, and EOT

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Clearview Cancer Institute Oncology Specialties, P.C, Huntsville, Alabama
  - University of Arizona SPORE, Tucson, Arizona
  - University of California San Diego, La Jolla, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Northwestern University, Chicago, Illinois
  - Horizon Oncology Center, Lafayette, Indiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mount Sinai School of Medicine and Mount Sinai Graduate School of Biological Sciences, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Cleveland Clinic, Cleveland, Ohio
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - US Oncology, The Woodlands, Texas

REFERENCES:
- [Background] Arnason JE, Brown JR. B cell receptor pathway in chronic lymphocytic leukemia: specific role of CC-292. Immunotargets Ther. 2014 Jan 24;3:29-38. doi: 10.2147/ITT.S37419. eCollection 2014. PMID 27471698
- See also: Leukemia & Lymphoma Society — http://www.lls.org/